CLINICAL TRIAL: NCT00072956
Title: The Physiology of Tricks
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040041; 04-N-0041
Record Dates: First submitted 2003-11-12; First posted 2003-11-13 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Dystonia; Torticollis
Keywords: Transcranial Magnetic Stimulation; Torticollis; Cervical Dystonia; Surround Inhibition; Sensory Tricks
MeSH Terms: conditions — Dystonia; Torticollis

SUMMARY:
This study will examine the action of sensory tricks on an occurrence known as surround inhibition when there is a disorder of muscle tone affecting a single body part in isolation. Surround inhibition refers to a situation that suppresses unwanted movements, known as dystonia, in surrounding muscles during voluntary actions. There are tricks-various actions-that people use to temporarily stop those unwanted movements. Such tricks can include touching the affected body part, placing an object in the mouth, pulling the hair, and others. Often these tricks are beneficial early in the illness but become less effective as it progresses. This study is guided by a hypothesis that sensory tricks will restore surround inhibition and by another hypothesis that it is the application of the tricks, not simply sensory input, that is effective in doing that restoring. Emphasis is on cervical dystonia, involuntary actions affecting the neck, in which the tricks commonly involve the cheeks and chin. The technique used in the study is transcranial magnetic stimulation (TMS).

Patients ages 18 and older who have cervical dystonia with at least one effective trick and patients with no effective trick may be eligible for this study. There will also be a control group of healthy participants.

Participants will be asked to show the sensory trick and may be asked to be videotaped. During the TMS procedure, they will be seated in a comfortable chair, with hands placed on a pillow on the lap. Small electrodes-soft strips that stick to the skin-will be placed on the skin to record the electrical activity of some muscles in the neck that are activated by the stimulation from TMS. In TMS, there will be a wire coil held over the scalp. A brief electrical current will be passed through the coil, creating a magnetic pulse that stimulates the brain. Patients will hear a click and may feel a pulling sensation on the skin under the coil. There may be muscle twitches of the face, arm, or leg. In addition, patients may be asked to tense certain muscles slightly or perform other simple actions so that the coil can be positioned appropriately. Patients will sometimes be asked to bite down and tap their teeth slightly for about 1-1/2 minutes at a time. They will be asked to show the sensory trick. The stimulation is usually not painful, although sometimes strong contractions of the scalp muscles can cause discomfort or a headache. Patients can ask to have the procedure discontinued at any time. The testing session takes about 2 hours, done on an outpatient basis.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the mechanism of sensory tricks on surround inhibition in the motor cortex in focal dystonia. Sensory tricks or Geste antagoniste, are various manoeuvres used by dystonic patients to transiently diminish their spasms. Many of these manoeuvres involve motor as well as sensory input and here we use the term 'tricks' to refer to both phenomena. Little is known of this unique feature that is an evidence for the abnormality of sensorimotor integration in focal dystonia. The relief of dystonic symptoms by the application of tricks suggests its potential as a clue to the understanding of the yet unclear mechanism of dystonia. There is evidence that surround inhibition, a cortical phenomenon that functions to suppress unwanted movements in surrounding muscles during voluntary actions, is impaired in dystonia. Since tricks transiently relieve the dystonic symptoms, we hypothesize that the mechanism of tricks is the normalization of surround inhibition which is defective in dystonia.

ELIGIBILITY:
INCLUSION CRITERIA:

Nineteen patients age 18 or over with cervical dystonia with a minimal of one effective trick, 15 patients age 18 and over with cervical dystonia with no effective trick will be recruited for the study.

For patients, the selection criteria are the presence of cervical dystonia and the minimal of one sensory trick in the patient with trick group, and no trick in the patient without trick group.

The interview of dystonic patients will be focused on medical history, neurologic examination and effectiveness of the patient's tricks which will be accessed by measuring the degree of head rotation before and during trick application.

The diagnosis of dystonia will rely on review of medical record, history, and clinical evaluation.

For the patients that are receiving botulinum toxin injections, the evaluation will be done 3 months after their last injection.

Their gender, age, or ethnic origin will not provide bias for inclusion to the study.

There is no evidence of higher prevalence of dystonia in any particular race, thus the races and ethnicity of the subjects recruited for this study will approximate that of the general population.

Fifteen normal subjects age 18 and over will be recruited for the control group.

The controls will not have dystonia or any other neurological condition.

All subjects will sign an informed consent prior to participation in the trial, and the trial will be approved by the NINDS IRB committee.

EXCLUSION CRITERIA:

Exclusion criteria for the trial covering both the normal control and dystonia group will include;

1. Any concurrent medical or surgical condition as well as neurological or psychiatric illnesses.
2. Any individual who is on medications with potential influence of the nervous system function (antidepressants, antianxiolytics, anticonvulsants, antipsychotic, antiparkinsonian, hypnotics, and stimulants).
3. Patients who have received Botulinum toxin injections within 3 months of starting the protocol.
4. Individual who has a pacemaker, an implanted medical pump, a metal plate or medical object in the skull or eye (for example, after brain surgery)
5. Individual with a history of seizures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49
Dates: Start 2003-11; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Abbruzzese G, Marchese R, Buccolieri A, Gasparetto B, Trompetto C. Abnormalities of sensorimotor integration in focal dystonia: a transcranial magnetic stimulation study. Brain. 2001 Mar;124(Pt 3):537-45. doi: 10.1093/brain/124.3.537. PMID 11222454
- [Background] Bara-Jimenez W, Shelton P, Sanger TD, Hallett M. Sensory discrimination capabilities in patients with focal hand dystonia. Ann Neurol. 2000 Mar;47(3):377-80. PMID 10716260
- [Background] Berardelli A, Rothwell JC, Hallett M, Thompson PD, Manfredi M, Marsden CD. The pathophysiology of primary dystonia. Brain. 1998 Jul;121 ( Pt 7):1195-212. doi: 10.1093/brain/121.7.1195. PMID 9679773